CLINICAL TRIAL: NCT04725864
Title: Vaginal Progesterone as Luteal Support for Improvement of Live Birth in Frozen/Thawed In-vitro Fertilization Natural Cycles; a Multicenter, Open, Randomized Trial
Brief Title: Progesterone as Luteal Support in Frozen IVF Natural Cycles
Acronym: ProFET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-005552-38
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Infertility; Embryo Transfer
Keywords: progesterone; luteal phase support; frozen embryo transfer; natural cycles; live birth
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Two main arms, of which the experimental arm is split in two arms with different duration of treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No progesterone (No Intervention): Patients will have FET in natural cycles with no extra intervention.
- Progesterone for 3 weeks (Experimental): At day LH+3 patients will start treatment with vaginal progesterone tablet at 100mg three times daily for three weeks.
  Interventions: Drug: Progesterone vaginal tablet
- Progesterone for 7 weeks (Experimental): At day LH+3 patients will start treatment with vaginal progesterone tablet at 100mg three times daily for seven weeks.
  Interventions: Drug: Progesterone vaginal tablet

INTERVENTIONS:
Drug: Progesterone vaginal tablet — The study drug is progesterone 100 mg administrated as a vaginal tablet three times daily.
  Other Names: Lutinus, manufactured by Ferring GmbH. ATC code G03DA04
  Arms: Progesterone for 3 weeks; Progesterone for 7 weeks

SUMMARY:
The ProFET study aims to investigate if luteal phase support by vaginal progesterone, is superior to no luteal phase support, in terms of live birth rate per woman after a frozen embryo transfer (FET), in a natural cycle (NC) after in-vitro fertilization (IVF), and if 7 weeks of treatment is superior to 3 weeks duration.

DETAILED DESCRIPTION:
Vaginal progesterone supplementation is routine treatment after IVF with fresh embryo transfer, but it is uncertain whether vaginal progesterone after frozen embryo transfer in natural cycles is efficacious in terms of increasing the chance of a live birth.

The ProFET study is a multicenter, open randomized, controlled trial planning to include 1800 women, intended to undergo a FET in a natural cycle.

Primary objectives are to investigate if luteal phase support by vaginal progesterone, is superior to no luteal phase support, in terms of live birth rate per woman after a frozen embryo transfer, in a natural cycle and if 7 weeks of treatment is superior to 3 weeks duration.

Secondary objectives are to compare groups regarding pregnancy outcomes including biochemical pregnancy, clinical, ongoing and term pregnancy rates, as well as rates of miscarriage, termination of pregnancy, and ectopic pregnancy.

Secondary objectives are also perinatal and obstetrics outcomes, self-reported side effects, adverse events and cost effectiveness.

The investigators will also analyze the effect of S-Progesterone level before FET on the chance of achieving live birth and secondary pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Planned for a FET-NC with a blastocyst
* BMI >18.5 <35
* Regular menstrual cycles 24-35 days
* Given informed consent
* Understand written and spoken Swedish, English or Arabic

Exclusion Criteria:

* Oocyte donor cycles, preimplantation genetic testing (PGT) cycles. Uterine malformation, submucous myoma and endometrial polyps.
* Hypersensitivity against study medication. Other contraindications according to www.fass.se
* Development of serious disease contraindicating ART or pregnancy.
* Participation or recent participation in a clinical study with an investigational product (past 30 days). Previous participation in this study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with live birth | Up to 41 weeks after embryo transfer.
  A child born alive. Also, the outcome will be reported according to Core Outcome Measure for Infertility Trials (Duffy et al., 2020) in a separate appendix.

SECONDARY OUTCOMES:
Number of participants with biochemical pregnancy | 2-3 weeks after embryo transfer.
  A pregnancy diagnosed only by the detection of beta hCG in serum or urine.
Number of participants with clinical pregnancy | 4-8 weeks after embryo transfer.
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs.
Number of participants with ongoing pregnancy | 5-7 weeks after embryo transfer.
  An intrauterine pregnancy with one or more fetuses with heartbeats measured in gestational week 7+5 to 9+0 with vaginal ultrasound.
Number of participants with miscarriage | Up to 20 weeks after embryo transfer.
  The spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age. Also, the outcome will be reported according to Core Outcome Measure for Infertility Trials (Duffy et al., 2020) in a separate appendix.
Number of participants with ectopic pregnancy | Up to 20 weeks after embryo transfer.
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Number of participants with termination of pregnancy | Up to 20 weeks after embryo transfer.
  Defined as the termination of a clinical pregnancy, by deliberate interference that takes place before 22 completed weeks of gestational age. Also, the outcome will be reported according to Core Outcome Measure for Infertility Trials (Duffy et al., 2020) in a separate appendix.
Birth weight | Up to 41 weeks after embryo transfer.
  Defined as weight in grams at birth.
Gestational age at delivery | Up to 41 weeks after embryo transfer.
  The gestational age at FET is calculated by adding the number of culture days to ovulation (ovulation=day 14). Gestational age at delivery is then calculated by adding the number of days since FET.
Preterm birth | Up to 35 weeks after embryo transfer.
  Defined as a child born alive before 37 completed weeks of pregnancy.
Very preterm birth | Up to 30 weeks after embryo transfer.
  Defined as a child born alive before 32 completed weeks of pregnancy.
Low birth weight | Up to 41 weeks after embryo transfer.
  Birth weight less than 2500 g.
Very low birth weight | Up to 41 weeks after embryo transfer.
  Birth weight less than 1500 g.
Stillbirth | Up to 41 weeks after embryo transfer.
  The death of a fetus prior to the complete expulsion or extraction from its mother, after and including 22 completed weeks of gestational age. Also, the outcome will be reported according to Core Outcome Measure for Infertility Trials (Duffy et al., 2020) in a separate appendix.
Perinatal death | Up to 41 weeks after embryo transfer and 7 days after birth.
  Fetal or neonatal death occurring during late pregnancy (at 22 completed weeks of gestational age and later), during childbirth, or up to seven days after birth. Also, the outcome will be reported according to Core Outcome Measure for Infertility Trials (Duffy et al., 2020) in a separate appendix.
Number of children with birth defects | Up to 41 weeks after embryo transfer.
  Congenital birth defects were defined according the International Statistical Classification of Diseases and Related Health Problems (ICD-10). And further defined according to the EUROCAT classification system.
Number of children admitted to Neonatal Intensive Care Unit (NICU) | Up to 41 weeks after embryo transfer and 7 days after birth.
  Defined as children that were admitted to NICU after birth.
Number of participants with hypertensive disorders of pregnancy | Up to 41 weeks after embryo transfer including the postpartum period before discharge of mother.
  Hypertensive disorders of pregnancy defined as high blood pressure disorders including preeclampsia, gestational hypertension and chronic hypertension.
Number of participants with placenta previa | Up to 41 weeks after embryo transfer.
  Defined as a placenta covering the internal os of the cervix, at time of delivery.
Number of participants with placenta abruption | Up to 41 weeks after embryo transfer.
  Defined as the premature separation of a normally located placenta from the uterine wall that occurs before delivery of the fetus.
Number of participants with postpartum hemorrhage | Up to 41 weeks after embryo transfer.
  Defined as a cumulative blood loss of greater than 1,000 mL or blood loss accompanied by signs or symptoms of hypovolemia within 24 hours after the birth process.
Number of participants with Cesarean section | Up to 41 weeks after embryo transfer.
  Defined as a surgical procedure used to deliver a baby through incisions in the abdomen and uterus.
Number of participants with thromboembolic events | Up to 41 weeks after embryo transfer including the postpartum period before discharge of mother.
  Defined as formation in a blood vessel of a clot (thrombus) that breaks loose and is carried by the blood stream to plug another vessel.
Maternal mortality | Up to 41 weeks after embryo transfer including the postpartum period before discharge of mother.
  Defined as female deaths from any cause related to or aggravated by pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth.
Number of participants with treatment related side effects | Up to 8 weeks after embryo transfer.
  Side effects reported according to study specific questionnaire. Questions are answered with yes or no. If yes, symptoms are described, but not by using a scale.
Number of participants with adverse events | Up to 8 weeks after embryo transfer.
  Any untoward medical occurrence in symptom or disease temporally associated with the use of the medicinal (investigational) product, whether or not related to the medicinal product.
Cost effectiveness | After study completion, an average of 1 year.
  Comparison between groups regarding the total costs for the intervention divided by treatment efficacy (live birth).

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Magnusson, MD, PhD, Principal Investigator — Vastra Gotaland
Locations (1):
- Department of Reproductive Medicine, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duffy JMN, AlAhwany H, Bhattacharya S, Collura B, Curtis C, Evers JLH, Farquharson RG, Franik S, Giudice LC, Khalaf Y, Knijnenburg JML, Leeners B, Legro RS, Lensen S, Vazquez-Niebla JC, Mavrelos D, Mol BWJ, Niederberger C, Ng EHY, Otter AS, Puscasiu L, Rautakallio-Hokkanen S, Repping S, Sarris I, Simpson JL, Strandell A, Strawbridge C, Torrance HL, Vail A, van Wely M, Vercoe MA, Vuong NL, Wang AY, Wang R, Wilkinson J, Youssef MA, Farquhar CM; Core Outcome Measure for Infertility Trials (COMMIT) initiative. Developing a core outcome set for future infertility research: an international consensus development studydagger double dagger. Hum Reprod. 2020 Dec 1;35(12):2725-2734. doi: 10.1093/humrep/deaa241. PMID 33252685
- [Derived] Stadelmann C, Bergh C, Brannstrom M, Olsen KH, Khatibi A, Kitlinski M, Liffner S, Lundborg E, Rodriguez-Wallberg KA, Strandell A, Westlander G, Widlund G, Magnusson A. Vaginal progesterone as luteal phase support in natural cycle frozen-thawed embryo transfer (ProFET): protocol for a multicentre, open-label, randomised controlled trial. BMJ Open. 2022 Jul 8;12(7):e062400. doi: 10.1136/bmjopen-2022-062400. PMID 35803628
- See also: EUROCAT classification system — https://eu-rd-platform.jrc.ec.europa.eu/sites/default/files/Full_Guide_1_4_version_28_DEC2018.pdf